# **Clinical Study Protocol**

## Retrospective clinical evaluation of nano-hybridcomposite denture teeth SR Phonares II

| Type of investigation: | Clinical investigation concerning medical devices | |
|---|---|---|
| Categorisation: | Category according to Art 6 ClinO-MD: A1 | |
| Registration: | Registry at ClinicalTrials.gov of the U.S. National Library of Medicine (http://www.clinicaltrials.gov) | |
| | The trial additionally registers in the supplementary federal database (Portal for clinical trials in Switzerland - SNCTP, https://www.kofam.ch/en/snctp-portal/) with its submission on BASEC. | |
| | Furthermore, as soon as the new electronic system EUDAMED2 is operational, the clinical investigation will be retrospectively registered, if required. | |
| Identifier: | LL 5267725 | |
| Principal Investigator and<br>Sponsor, or Sponsor-<br>Investigator: | Principal Investigator (PI): Dr. med. dent. Ronny Watzke Bendererstrasse 2 9494 Schaan Fürstentum Liechtenstein Tel.: Mail: Sponsor: Ivoclar Vivadent AG Bendererstrasse 2 | |
| | 9494 Schaan | |
| | Fürstentum Liechtenstein | |
| Sponsor representative (if the Sponsor is not located in | Patrik Oehri | |
| Switzerland) | Senior Director Corporate Quality Management/PRRC | |
| | Tel.: Mail: | |
| Medical Device: | SR Phonares II (Ivoclar Vivadent AG) | |
| | Article | UDI |
| | SR Phonares II Ant. 6er OS71 A2 | DIVO6448651 |
| | SR Phonares II Ant. 6er OS71 A3 | DIVO6448661 |
| | SR Phonares II Ant. 6er OS72 A3 | DIVO6448861 |
| | SR Phonares II Ant. 6er OB71 A3 | DIVO6450461 |

LL 5267725 Version 2.0, 19.09.2022 

| | SR Phonares II Ant. 6er OB72 A3 | DIVO6450661 |
|-------------------|-----------------------------------|-------------|
| | SR Phonares II Ant. 6er OB73 A3 | DIVO6450861 |
| | SR Phonares II Ant. 6er OB73 A3.5 | DIVO6450871 |
| | SR Phonares II Ant. 6er UL50 A2 | DIVO6451651 |
| | SR Phonares II Ant. 6er UL51 A3 | DIVO6451861 |
| | SR Phonares II Ant. 6er UL51 A3.5 | DIVO6451871 |
| | SR Phonares II Ant. 6er UL52 A3 | DIVO6452061 |
| | SR Phonares II Ant. 6er UL53 A3 | DIVO6452261 |
| | SR Phonares II Typ 8er ONU3 A3 | DIVO6453661 |
| | SR Phonares II Typ 8er ONU5 A3 | DIVO6453861 |
| | SR Phonares II Typ 8er ONU5 A3.5 | DIVO6453871 |
| | SR Phonares II Typ 8er ONU6 A3 | DIVO6454061 |
| | SR Phonares II Typ 8er UNL3 A2 | DIVO6454251 |
| | SR Phonares II Typ 8er UNL5 A3 | DIVO6454461 |
| | SR Phonares II Typ 8er UNL5 A3.5 | DIVO6454471 |
| Version and Date: | Version 2.0, 19.09.2022 | |

#### CONFIDENTIAL

The information contained in this document is confidential and the property of the Ivoclar Vivadent AG. The information may not - in full or in part - be transmitted, reproduced, published, or disclosed to others than the applicable Competent Ethics Committee(s) and Regulatory Authority(ies) without prior written authorisation from the Sponsor except to the extent necessary to obtain informed consent from those who will participate in the investigation.

LL 5267725 Version 2.0, 19.09.2022 

#### Signature Page(s)

ID number of the

LL 5267725

investigation:

Registry at ClinicalTrials.gov of the U.S. National Library of

Medicine (http://www.clinicaltrials.gov):

The trial additionally registers in the supplementary federal database (Portal for clinical trials in Switzerland - SNCTP, https://www.kofam.ch/en/snctp-portal/) with its submission on

BASEC.

Furthermore, as soon as the new electronic system EUDAMED2 is operational, the clinical investigation will be retrospectively

registered, if required.

Title:

Retrospective clinical evaluation of nano-hybrid-composite

denture teeth SR Phonares II

The Sponsor, the Principal Investigator and the Statistician have approved the CIP version 1.0 (dated 23.08.2022) and confirm hereby to conduct the investigation according to the CIP, the current version of the World Medical Association Declaration of Helsinki, ISO14155 norm, ICH-GCP as far as applicable, and the local legally applicable requirements.

| Sponsor-Representative:<br>Patrik Oehri | |
|-----------------------------------------|-----------|
| Schaan, 19. 09. 2022 | |
| Place/Date | Signature |

Principal Investigator:

Dr. med. dent. Ronny Watzke

Signature

## 1. SYNOPSIS

| Sponsor / Sponsor-<br>Investigator | Ivoclar Vivadent AG |
|---|---|
| Title: | Retrospective clinical evaluation of nano-hybrid-composite denture teeth SR Phonares II |
| Short title / | Retrospective clinical evaluation of SR Phonares II |
| Investigation ID: | Investigation ID: LL 5267725 |
| Clinical Investigation Plan, version and date: | Version 2.0, 19.09.2022 |
| Registration: | Registry at ClinicalTrials.gov of the U.S. National Library of Medicine (http://www.clinicaltrials.gov): |
| | The trial additionally registers in the supplementary federal database (Portal for clinical trials in Switzerland - SNCTP, https://www.kofam.ch/en/snctp-portal/) with its submission on BASEC. |
| | Furthermore, as soon as the new electronic system EUDAMED2 is operational, the clinical investigation will be retrospectively registered, if required. |
| Category and its | Category A1 |
| rationale: | The medical device has conformity marking and will be used according to its instruction for use. The subjects are not subjected to any additional invasive or stressful procedures compared with those applied under normal conditions of use of the product. |

LL 5267725 Version 2.0, 19.09.2022 

| Name of the MD, | SR Phonares II | |
|---|---|---|
| Unique Device | | |
| Identification (UDI), name of the | Article UDI | |
| manufacturer | SR Phonares II Ant. 6er OS71 A2 DIVO6448651 | |
| | SR Phonares II Ant. 6er OS71 A3 | DIVO6448661 |
| | SR Phonares II Ant. 6er OS72 A3 | DIVO6448861 |
| | SR Phonares II Ant. 6er OB71 A3 | DIVO6450461 |
| | SR Phonares II Ant. 6er OB72 A3 | DIVO6450661 |
| | SR Phonares II Ant. 6er OB73 A3 | DIVO6450861 |
| | SR Phonares II Ant. 6er OB73 A3.5 | DIVO6450871 |
| | SR Phonares II Ant. 6er UL50 A2 | DIVO6451651 |
| | SR Phonares II Ant. 6er UL51 A3 | DIVO6451861 |
| | SR Phonares II Ant. 6er UL51 A3.5 | DIVO6451871 |
| | SR Phonares II Ant. 6er UL52 A3 | DIVO6452061 |
| | SR Phonares II Ant. 6er UL53 A3 | DIVO6452261 |
| | SR Phonares II Typ 8er ONU3 A3 | DIVO6453661 |
| | SR Phonares II Typ 8er ONU5 A3 | DIVO6453861 |
| | SR Phonares II Typ 8er ONU5 A3.5 | DIVO6453871 |
| | SR Phonares II Typ 8er ONU6 A3 | DIVO6454061 |
| | SR Phonares II Typ 8er UNL3 A2 | DIVO6454251 |
| | SR Phonares II Typ 8er UNL5 A3 | DIVO6454461 |
| | SR Phonares II Typ 8er UNL5 A3.5 | DIVO6454471 |
| | Ivoclar Vivadent AG | |
| | Benderer Strasse 2 | derer Strasse 2 |
| | 9494 Schaan | an |
| Stage of development: | Post-market stage with CE marking | |
| Background and rationale: | This retrospective study investigates the longevity of dentures with SR Phonares II teeth after a wearing period of more than 10 years. | |
| Objective(s): | The primary objective is to assess the survival rate of dentures with SR Phonares II teeth after more than 10 years. The secondary objectives asses the quality of the dentures concerning aesthetic, functional and biological properties. | |
| Outcome(s): | The primary outcome of the study is the survival rate of the dentures with the tested denture teeth. The secondary outcomes are all linked to the quality of the materials used (surface lustre, staining, plaque accumulation, color match, aesthetic anatomical form, fracture, marginal adaptation, occlusal contour, wear patients view, integrity of adjacent natural teeth, adjacent mucosa, oral health). | |
| Design: | Retrospective evaluation | |

LL 5267725 Version 2.0, 19.09.2022 

| Inclusion / exclusion criteria: | Subjects fulfilling all <u>inclusion</u> criteria are eligible for the investigation: informed consent signed and understood by the subject, partial or full denture with SR Phonares II teeth, dentures delivered in the internal clinic between August 2010 and August 2012, to be able to visit the internal clinic (Exception: Patients with limited mobility are also included if another person can carry the dentures to the internal clinic of Ivoclar Vivadent AG for the examination.). The presence of any of the following <u>exclusion</u> criteria will lead to the exclusion of the subject: patient does not wear the dentures regularly, health status (physical and mental) does not allow participation. |
|---|---|
| Measurements and procedures: | The intraoral situation will be examined similar to a standard dental examination. The dentures are then removed, cleaned and examined extraoral. Pictures and an impression of the dentures are taken. |
| Intervention: | The examinations do not differ from standard dental examinations. Impressions of the back teeth of the dentures are taken extraoral and stone casts are poured. They are used for analysis of wear and microscopical analysis. |
| Control intervention (if applicable): | n.a. |
| Number of subjects with rationale: | 22 patients that were supplied with dentures with SR Phonares II teeth (in total 43 dentures) in the internal clinic of Ivoclar Vivadent AG between August 2010 and August 2012. |
| Duration of the investigation: | 6 months |
| Investigation | October 2022 First- subject –In (planned) |
| schedule: | March 2023 Last- subject –Out (planned) |
| Investigator(s): | Dr. med. dent. Ronny Watzke |
| | Bendererstrasse 2<br>9494 Schaan |
| | Fürstentum Liechtenstein |
| | Tel.: |
| | Mail: |
| Investigational | This is a single centre study. |
| Site(s): | R&D Clinic |
| | Ivoclar Vivadent AG |
| | Bendererstrasse 2 |
| | 9494 Schaan |
| | Fürstentum Liechtenstein |
| Statistical considerations: | Since the study is retrospective with a small cohort and no control group, mainly descriptive statistical analysis will be performed. The obtained data, especially the survival rate will be discussed and compared with data from the literature. A minimal sample size of 41 dentures was calculated with absolute error (precision of 10% and and standard normal variate of 5% (type 1 error)). |
| Compliance statement: | This investigation will be conducted in compliance with the CIP, the current version of the Declaration of Helsinki, ISO14155, ICH-GCP (as far as applicable) as well as all national legal and regulatory requirements. |

LL 5267725 Version 2.0, 19.09.2022 

#### 2. ABBREVIATIONS

AE Adverse Event

ADE Adverse Device Effect

ASADE Anticipated Serious Adverse Device Effect

ASR Annual Safety Report

CA Competent Authority (e.g. Swissmedic)

CEC Competent Ethics Committee
CIP Clinical investigation plan

ClinO Ordinance on Clinical Trials in Human Research (in German KlinV, in French Oclin,

in Italian OSRUm)

ClinO-MD Ordinance on Clinical Trials with Medical Devices (in German: KlinV-Mep, in French:

Oclin-Dim, in Italian: OSRUm-Dmed)

CRF Case Report Form (pCRF paper CRF; eCRF electronic CRF)

DD Device Deficiency

DMC / DSMC Data Monitoring Committee, Data Safety Monitoring Committee

Ho Null hypothesis

H1 Alternative hypothesis

HRA Federal Act on Research involving Human Beings (in German: HFG, in French:

LRH, in Italian: LRUm)

IB Investigator's Brochure
ICF Informed Consent Form

ICH-GCP International Council for Harmonisation – guidelines of Good Clinical Practice

IFU Instruction For Use ISF Investigator Site File

ISO International Organisation for Standardisation

ITT Intention to treat

MedDO Medical Devices Ordinance (in German: MepV, in French: Odim, in Italian: Odmed)

MD Medical Device

MDR Medical Device Regulation (EU) 2017/745 of 5 April 2017

PI Principal Investigator

SADE Serious Adverse Device Effect

SAE Serious Adverse Event SDV Source Data Verification

SNCTP Swiss National Clinical Trials Portal

SOP Standard Operating Procedure

USADE Unanticipated Serious Adverse Device Effect

LL 5267725 Version 2.0, 19.09.2022 

## 3. SUMMARY OF THE REVISION HISTORY IN CASE OF AMENDMENTS

| Version Nr,<br>Version Date | Chapter | Description of change | Reason for the change |
|---|---|---|---|

## 4. INVESTIGATION SCHEDULE

| Investigation Periods | Patient information | Consent (ICF) | Recall |
|------------------------------|---------------------|---------------|--------|
| Visit | 0 | 1 | 1 |
| Time (day) | -3 | 0 | 0 |
| Patient Information by phone | x | | |
| Patient consent (ICF) | | х | |
| Primary Variables | | | х |
| Secondary Variables | | | х |
| Dental radiograph | | | (x) |
| Adverse events | | | х |
| Device Deficiencies | | | х |

<sup>(</sup>x) dental radiographs of a single tooth or dental implant will only be taken if necessary for medical reasons independent of the clinical trial.

LL 5267725 Version 2.0, 19.09.2022 